CLINICAL TRIAL: NCT04750317
Title: Efficacy and Safety of Tofacitinib in Patients With COVID-19 Pneumonia
Acronym: TOFA-COV-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107892
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with reduced oxygen saturation ≤93% treated with tofacitinib (Experimental): Patients with oxygen saturation ≤93% on admission treated with tofacitinib and standard of care treatment
  Interventions: Drug: Tofacitinib
- Patients with reduced oxygen saturation treated with SoC (No Intervention): Patients with oxygen saturation ≤93% on admission treated with standard of care only
- Patients with preserved oxygen saturation >93% on admission treated with tofacitinib (Experimental): Patients with oxygen saturation >93% on admission treated with tofacitinib and standard of care
  Interventions: Drug: Tofacitinib
- Patients with preserved oxygen saturation >93% on admission treated with SoC (No Intervention): Patients with oxygen saturation >93% on admission treated with standard of care only

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib was administered at a dose 10 mg twice daily on day 1, followed by 5 mg twice daily on day 2-5. The dosage was reduced up to 5 mg once daily in patients with moderate renal impairment or moderate hepatic impairment.
  Arms: Patients with preserved oxygen saturation >93% on admission treated with tofacitinib; Patients with reduced oxygen saturation ≤93% treated with tofacitinib

SUMMARY:
TOFA-COV-2 is a cohort study of the efficacy of tofacitinib in reducing the risk of mechanical ventilation and/or death in patients with moderately severe COVID-19 pneumonia who received standard of care treatment (SoC). The study population consists of adults (≥18 years) with COVID-19, who are admitted to the university hospitals and don't require invasive or noninvasive ventilation on admission. All patients are divided into four groups depending on nadir levels of oxygen saturation and therapy: (1) patients with oxygen saturation ≤93% who received tofacitinib and SoC, (2) patients with oxygen saturation ≤93% who received only SoC, (3) patients with oxygen saturation >93% who received tofacitinib and SoC, (4) patients with oxygen saturation >93% who received only SoC. The aim of the study is to test the hypothesis that addition of tofacitinib to SoC could reduce the risk of mechanical ventilation and/or death.

DETAILED DESCRIPTION:
TOFA-COV-2 is a cohort study that is conducted in the three clinics of the Sechenov University (Moscow, Russia) in patients with moderately severe COVID-19 pneumonia. A diagnosis of COVID-19 associated pneumonia suspected clinically was confirmed by polymerase chain reaction (PCR) and/or chest CT. In patients with inconclusive or negative results of PCR on nasopharyngeal swab, SARS-CoV-2 induced pneumonia was defined as an acute respiratory infection with typical CT findings (4 or 5 on CO-RADS scale) and no other obvious aetiology.

In order to be included in this study, patients must have COVID-19 pneumonia involving at least 25% of lung tissue in combination with at least one of the following: (1) oxygen saturation at rest ≤93% on ambient air, (2) increased C-reactive protein (CRP ≥50 mg/L) and/or (3) fever (≥38.0°C) that persisted for at least two days despite treatment with nonsteroidal antiinflammatory drugs or paracetamol. Exclusion criteria for the administration of tofacitinib were coexistent infection other than COVID-19; requirement for invasive mechanical ventilation; estimated glomerular filtration rate calculated using CKD-EPI formula ≤30 ml/min/1.73 m2; elevated ALT and/or AST levels more than 3 times the upper limit of normal; chronic use of glucocorticoids or immunosuppressive agents; and administration of interleukin-6 inhibitors and/or high-dose glucocorticoids (≥250 mg prednisone equivalent intravenously) for the treatment of COVID-19.

All patients are divided into four groups depending on nadir levels of oxygen saturation and therapy: (1) patients with oxygen saturation ≤93% who received tofacitinib and SoC, (2) patients with oxygen saturation ≤93% who received only SoC, (3) patients with oxygen saturation >93% who received tofacitinib and SoC, (4) patients with oxygen saturation >93% who received only SoC. The aim of the study is to test the hypothesis that administration of tofacitinib could influence the risk of mechanical ventilation and/or death.

All patients provided written, informed consent for the off-label use of experimental medications, including tofacitinib, according to the provisional recommendations issued by the Russian Ministry of Health during the outbreak of infection.

ELIGIBILITY:
Inclusion Criteria:

1. SARS-CoV2 Infection diagnosed by PCR and/or typical lesions on CT-scan (4 or 5 on CO-RADS scale) in combination with at least one of the following:

   * oxygen saturation at rest ≤93% on ambient air,
   * AND/OR C-reactive protein ≥50 mg/L,
   * AND/OR fever (≥38.0°C) that persisted for at least two days despite treatment with nonsteroidal antiinflammatory drugs or paracetamol
2. Written Informed Consent

Exclusion Criteria:

1. Age <18 years
2. Coexistent infection other than COVID-19
3. Requirement for invasive mechanical ventilation
4. Estimated glomerular filtration rate calculated using CKD-EPI formula ≤30 ml/min/1.73 m2;
5. Elevated ALT and/or AST levels more than 3 times the upper limit of normal
6. Chronic use of glucocorticoids or immunosuppressive agents
7. Administration of interleukin-6 inhibitors and/or high-dose glucocorticoids (≥250 mg prednisone equivalent intravenously) for the treatment of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Death | Within 28 days from admission
  Death registered by medical personnel during in-hospital stay
Mechanical ventilation | Within 28 days from admission
  Initiation of mechanical ventilation during in-hospital stay in patients who did not require ventilation on admission

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Moiseev, MD, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Sechenov First Moscow State Medical University (Sechenov University) - University Clinical Hospital, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No